CLINICAL TRIAL: NCT07331701
Title: Association of BAL Fluid T-Cell Immune Activity With Tumor PD-L1 Expression and Its Prognostic Value: A Prospective Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Deog Kyeom Kim, Professor, Department of Pulmonary and Critical Care Medicine, SMG-SNU Boramae Medical Center, Seoul National University Hospital
Other Study IDs: BRMH 30-2025-48
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasms; Tumor Immune Microenvironment
Keywords: Bronchoalveolar Lavage Fluid; Tumor-Infiltrating T Lymphocytes; Programmed Cell Death 1 Ligand 1; Immune Checkpoint Inhibitors; Flow Cytometry; Tumor Immune Microenvironment; Treatment Response; Progression-Free Survival; Overall Survival; Predictive Biomarkers
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Lung Cancer Cohort: Adults with suspected or confirmed stage IV lung cancer undergoing clinically indicated bronchoscopy with bronchoalveolar lavage. Participants are enrolled prospectively as a single observational cohort, and no treatment assignment or intervention is determined by the study. Bronchoalveolar lavage fluid is collected for immune profiling by flow cytometry, and study analyses stratify participants post hoc according to tumor PD-L1 expression levels and bronchoalveolar lavage T-cell immunophenotypes.

SUMMARY:
This prospective observational study aims to evaluate whether immune profiles of T-cell subsets in bronchoalveolar lavage fluid can complement tumor PD-L1 expression, assessed by immunohistochemistry in tumor tissue specimens, in predicting clinical outcomes in patients with advanced lung cancer. Although tumor PD-L1 expression measured on tissue biopsies is widely used to guide immunotherapy decisions, its predictive value is limited by spatial heterogeneity and sampling variability. By analyzing activated, exhausted, and regulatory T-cell populations in bronchoalveolar lavage fluid and examining their association with tissue-based tumor PD-L1 expression, this study seeks to determine whether combining local immune biomarkers with PD-L1 expression improves the prediction of treatment response and survival in patients receiving standard-of-care systemic therapy.

DETAILED DESCRIPTION:
Tumor PD-L1 expression assessed by immunohistochemistry on tumor tissue specimens is an established biomarker for selecting immune checkpoint inhibitor therapy in lung cancer; however, its clinical utility is limited by intratumoral heterogeneity, temporal variability, and dependence on the size and location of tissue biopsy samples. As a result, tissue-based PD-L1 expression alone does not fully capture the immune context of the tumor microenvironment or reliably predict treatment response and prognosis in all patients.

Bronchoalveolar lavage fluid provides access to the local pulmonary immune microenvironment and contains immune cells that may reflect tumor-immune interactions more directly than peripheral blood. Prior studies suggest that T-cell populations in bronchoalveolar lavage fluid share phenotypic characteristics with tumor-infiltrating lymphocytes and may serve as surrogate indicators of local antitumor immune activity. However, the relationship between bronchoalveolar lavage T-cell immunophenotypes, tissue-based tumor PD-L1 expression, and clinical outcomes has not been comprehensively evaluated in a prospective setting.

This single-center prospective observational cohort study enrolls adult patients with suspected or confirmed stage IV lung cancer who are undergoing clinically indicated bronchoscopy as part of routine diagnostic or management procedures. Residual bronchoalveolar lavage fluid obtained during standard-of-care bronchoscopy is analyzed using multicolor flow cytometry to quantify T-cell subsets, including activated, exhausted, and regulatory populations defined by surface marker expression. Tumor PD-L1 expression is evaluated by immunohistochemistry performed on diagnostic tumor tissue specimens obtained as part of routine clinical care and analyzed both as a continuous variable and by predefined expression categories.

Participants receive standard systemic anticancer therapy according to current clinical guidelines, including immune checkpoint inhibitor-based regimens when indicated. Clinical outcomes, including objective response rate, progression-free survival, and overall survival, are prospectively collected from electronic medical records. The study examines correlations between bronchoalveolar lavage T-cell immunophenotypes and tissue-based tumor PD-L1 expression, as well as whether stratification based on combined immune profiling provides improved prognostic information compared with tumor PD-L1 expression alone.

By integrating local immune profiling from bronchoalveolar lavage fluid with tumor PD-L1 expression assessed in tissue specimens, this study seeks to identify complementary biomarkers that may enhance risk stratification and refine prognostic assessment in advanced lung cancer, potentially informing future approaches to personalized immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Patients with suspected or histologically confirmed stage IV lung cancer based on clinical and radiologic findings
* Scheduled to undergo clinically indicated bronchoscopy with bronchoalveolar lavage as part of routine clinical care
* Able and willing to provide written informed consent

Exclusion Criteria:

* Receipt of treatment for acute lower respiratory tract infection (including pneumonia or fungal infection) within 4 weeks prior to bronchoscopy
* History of solid organ transplantation or hematopoietic stem cell transplantation
* Current use of systemic immunosuppressive therapy
* Current or planned use of biologic immunomodulatory agents
* Known autoimmune disease requiring systemic immunosuppressive treatment
* Pregnant women
* Patients with recurrent stage IV lung cancer after prior definitive therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult patients evaluated at SMG-SNU Boramae Medical Center in Seoul, Republic of Korea. Participants are drawn from routine clinical practice and include patients undergoing clinically indicated bronchoscopy as part of the diagnostic evaluation or management of suspected or confirmed stage IV lung cancer. All clinical assessments, treatments, and follow-up are performed according to standard-of-care practice based on current clinical guidelines, and no additional diagnostic or therapeutic procedures are introduced solely for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Bronchoalveolar Lavage T-cell Immunophenotypes and Tumor PD-L1 Expression | At baseline, prior to initiation of systemic anticancer therapy
  The primary outcome is the association between T-cell immunophenotypes quantified in bronchoalveolar lavage fluid by multicolor flow cytometry and tumor PD-L1 expression assessed by immunohistochemistry. T-cell subsets include activated, exhausted, and regulatory T-cell populations defined by surface marker expression (e.g., PD-1, TIM-3, CD39, CD28, CD25, and CD127). Tumor PD-L1 expression is evaluated as the percentage of PD-L1-positive tumor cells and analyzed as a continuous variable and by predefined categories (<1%, 1-49%, ≥50%).

SECONDARY OUTCOMES:
Differences in Bronchoalveolar Lavage T-cell Immunophenotypes Across Tumor PD-L1 Expression Categories | At baseline, prior to initiation of systemic anticancer therapy
  This outcome compares bronchoalveolar lavage T-cell subset distributions among participants stratified by tumor PD-L1 expression categories (<1%, 1-49%, and ≥50%). T-cell immunophenotypes are assessed by flow cytometry and include proportions of activated, exhausted, and regulatory T-cell subsets.
Objective Response Rate by Combined Tumor PD-L1 Expression and Bronchoalveolar Lavage T-cell Immunophenotypes | From treatment initiation to first radiologic response assessment (typically 6-12 weeks)
  Objective response rate is defined as the proportion of participants achieving complete or partial response according to RECIST version 1.1. Objective response rates are evaluated using combined stratification by tumor PD-L1 expression categories and bronchoalveolar lavage T-cell immunophenotype profiles, and compared with response rates stratified by tumor PD-L1 expression alone to assess improvement in treatment response prediction.
Progression-Free Survival by Combined Tumor PD-L1 Expression and Bronchoalveolar Lavage T-cell Immunophenotypes | From treatment initiation to disease progression or death, up to approximately 24 months
  Progression-free survival is defined as the time from initiation of systemic anticancer therapy to disease progression or death from any cause, whichever occurs first. Progression-free survival is analyzed using combined stratification based on tumor PD-L1 expression categories (<1%, 1-49%, ≥50%) and bronchoalveolar lavage T-cell immunophenotype profiles. Survival outcomes using the combined stratification are compared with those based on tumor PD-L1 expression categories alone to evaluate the incremental prognostic value of bronchoalveolar lavage immune profiling.
Overall Survival by Combined Tumor PD-L1 Expression and Bronchoalveolar Lavage T-cell Immunophenotypes | From treatment initiation to death from any cause, up to approximately 24 months
  Overall survival is defined as the time from initiation of systemic anticancer therapy to death from any cause. Overall survival is analyzed according to combined stratification by tumor PD-L1 expression categories and bronchoalveolar lavage T-cell immunophenotype profiles. Survival outcomes derived from the combined model are compared with those based on tumor PD-L1 expression alone to assess whether bronchoalveolar lavage immune profiling improves prognostic discrimination.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, Dongjak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. The study includes sensitive clinical, immunologic, and imaging data derived from bronchoalveolar lavage samples and other patient-specific assessments, and no formal data-sharing infrastructure or governance plan has been established at the time of trial registration. However, de-identified individual participant data that underlie the results reported in peer-reviewed publications may be made available after publication upon reasonable request to the corresponding author, subject to appropriate data use agreements, institutional approval, and compliance with applicable ethical and privacy regulations.

REFERENCES:
- [Result] Kim IA, Hur JY, Kim HJ, Kim WS, Lee KY. Extracellular Vesicle-Based Bronchoalveolar Lavage Fluid Liquid Biopsy for EGFR Mutation Testing in Advanced Non-Squamous NSCLC. Cancers (Basel). 2022 May 31;14(11):2744. doi: 10.3390/cancers14112744. PMID 35681723
- [Result] Kalkanis A, Papadopoulos D, Testelmans D, Kopitopoulou A, Boeykens E, Wauters E. Bronchoalveolar Lavage Fluid-Isolated Biomarkers for the Diagnostic and Prognostic Assessment of Lung Cancer. Diagnostics (Basel). 2022 Nov 25;12(12):2949. doi: 10.3390/diagnostics12122949. PMID 36552956
- [Result] Masuhiro K, Tamiya M, Fujimoto K, Koyama S, Naito Y, Osa A, Hirai T, Suzuki H, Okamoto N, Shiroyama T, Nishino K, Adachi Y, Nii T, Kinugasa-Katayama Y, Kajihara A, Morita T, Imoto S, Uematsu S, Irie T, Okuzaki D, Aoshi T, Takeda Y, Kumagai T, Hirashima T, Kumanogoh A. Bronchoalveolar lavage fluid reveals factors contributing to the efficacy of PD-1 blockade in lung cancer. JCI Insight. 2022 May 9;7(9):e157915. doi: 10.1172/jci.insight.157915. PMID 35389889
- [Result] Mariniello A, Tabbo F, Indellicati D, Tesauro M, Rezmives NA, Reale ML, Listi A, Capelletto E, Carnio S, Bertaglia V, Mecca C, Consito L, De Filippis M, Bungaro M, Paratore C, Di Maio M, Passiglia F, Righi L, Sangiolo D, Novello S, Geuna M, Bironzo P. Comparing T Cell Subsets in Broncho-Alveolar Lavage (BAL) and Peripheral Blood in Patients with Advanced Lung Cancer. Cells. 2022 Oct 14;11(20):3226. doi: 10.3390/cells11203226. PMID 36291098
- [Result] Mansour MSI, Hejny K, Johansson F, Mufti J, Vidis A, Mager U, Dejmek A, Seidal T, Brunnstrom H. Factors Influencing Concordance of PD-L1 Expression between Biopsies and Cytological Specimens in Non-Small Cell Lung Cancer. Diagnostics (Basel). 2021 Oct 18;11(10):1927. doi: 10.3390/diagnostics11101927. PMID 34679625
- [Result] Ben Dori S, Aizic A, Sabo E, Hershkovitz D. Spatial heterogeneity of PD-L1 expression and the risk for misclassification of PD-L1 immunohistochemistry in non-small cell lung cancer. Lung Cancer. 2020 Sep;147:91-98. doi: 10.1016/j.lungcan.2020.07.012. Epub 2020 Jul 13. PMID 32683207
- [Result] Gniadek TJ, Li QK, Tully E, Chatterjee S, Nimmagadda S, Gabrielson E. Heterogeneous expression of PD-L1 in pulmonary squamous cell carcinoma and adenocarcinoma: implications for assessment by small biopsy. Mod Pathol. 2017 Apr;30(4):530-538. doi: 10.1038/modpathol.2016.213. Epub 2017 Jan 6. PMID 28059094